CLINICAL TRIAL: NCT03837769
Title: Single-center Intervention Study to Validate the Performance of the Aktiia SA PulseWatch Optical Blood Pressure Monitoring (OBPM) Device at the Wrist Against Invasive Blood Pressure Measurements With Arterial Line
Brief Title: Validation of the Aktiia SA PulseWatch OBPM Device at the Wrist Against Invasive Blood Pressure Measurements
Acronym: OBPM_ICU2018
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Neuchatelois (Other)
Collaborators: Aktiia SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: OBPM_ICU2018
Record Dates: First submitted 2019-02-06; First posted 2019-02-12 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Blood Pressure
Keywords: Blood Pressure; OBPM; Cuffless

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aktiia SA PulseWatch (Experimental): Aktiia OBPM PulseWatch wrist device
  Interventions: Device: Aktiia OBPM PulseWatch wrist device

INTERVENTIONS:
Device: Aktiia OBPM PulseWatch wrist device — The optical signals at the wrist are recorded non-invasively. The BP measurements are further determined from these optical signals and are compared to the reference BP readings.

SUMMARY:
Single-centre intervention study to validate the performance of the Aktiia SA optical blood pressure monitoring (OBPM) device at the wrist against invasive blood pressure measurements with arterial line.

DETAILED DESCRIPTION:
Aktiia SA PulseWatch is an investigational device for the optical measurement of blood pressure that uses only optical sensors at the wrist. HNE is interested in exploring the potential of the device and technology (OBPM), and aims at benchmarking its performances against gold standard measurements of blood pressure.

The goal of this study is thus to assess whether i) PulseWatch allows to capture blood pressure variations, and ii) the measured blood pressure values remain stable in time.

The proposed study plans to include patients that are already scheduled for arterial catheterization at HNE. For these patients, the study will only require the placement of the safe optical device on the wrist to non-invasively record hemodynamic fluctuations. Therefore, no additional risk for the patient is to be foreseen.

By demonstrating that the Aktiia SA OBPM technology is reliable, HNE aims to make one step further in improving blood pressure monitoring in general, and in particular in advancing the deployment of technologies that have the potential to be used in the ambulatory setting. The diagnosis and treatment of hypertension are expected to largely benefit from these advancements.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* No significant non-invasive systolic blood pressure difference between left arm and right arm (difference <20mmHg in systolic arterial pressure)
* Patient requires continuous monitoring of diastolic and systolic blood pressure continuously via a radial arterial line;
* Patient information and informed consent is obtained following the procedures described in CIP

Exclusion criteria:

* Arrythmias: tachycardia (resting heart rate > 120/min) at time of study inclusion
* Atrial fibrillation
* Psychomotor agitation
* Significant bruises or trauma on forearm
* Intravenous canula around the wrist with impossibility to place the device (Aktiia OBPM PulseWatch) around the wrist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-05-22 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Cuffless Blood Pressure performance | 4 Months
  The evaluation of the accuracy (mean error and standard deviation of the error) of the non-invasive BP measurements at wrist with the PulseWatch against the reference gold-standard invasive blood pressure obtained by arterial line with respect to ISO 81060-2 (14) for two aspects: i) capturing the variations of the BP in short time and ii) maintaining the accurate stable measurements over extended periods of time.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital neuchâtelois - Pourtalès, Neuchâtel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aktiia SA website — http://www.aktiia.com